CLINICAL TRIAL: NCT00027183
Title: Role of Exotoxins in the Pathogenesis of Pseudomonas Aeruginosa
Brief Title: Role of Toxins in Lung Infections Caused by Pseudomonas Aeruginosa
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980062; 98-H-0062
Record Dates: First submitted 2001-11-27; First posted 2001-11-28 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Pseudomonas Infection; Cystic Fibrosis
Keywords: Cystic Fibrosis; Effector Proteins; Cytotoxin; Lung Injury; Genetic Screen; Natural History
MeSH Terms: conditions — Pseudomonas Infections; Cystic Fibrosis; Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Healthy Volunteers
- 2: Cystic Fibrosis subjects

SUMMARY:
Some bacteria that cause disease can produce toxic substances that may worsen the disease. Pseudomonas aeruginosa is a bacteria that can produce a variety of toxins and is of special interest for patients with cystic fibrosis and repeated long term lung infections.

The goal of this study is to determine whether specific toxins produced by Pseudomonas aeruginosa may be important in the disease process of chronic lung infections of patients with cystic fibrosis.

This study will attempt to measure bacterial production of toxins in blood and sputum and immune system response to toxins in the blood....

DETAILED DESCRIPTION:
The goal of this study is to determine whether virulence determinants that use the type III-secretory pathway may be important in the pathogenesis of chronic Pseudomonas aeruginosa lung infections in patients with cystic fibrosis (CF). The studies will quantify bacterial effector proteins in serum and sputum and the immune response to specific products as reflected by antibodies in serum. Candidate effector proteins include: (1) exotoxin A, a non-type III-dependent ADP-ribosyltransferase and cytotoxin that does not use the Type III secretory pathway, (2) ExoS, a type III pathway-dependent extracellular ADP-ribosyltransferase with cytotoxic activity, (3) ExoU, another type III-dependent cytotoxin, that is responsible for epithelial injury in acute lung infections, and (4) PcrV, a homolog to the V antigen of Yersinia.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with cystic fibrosis with a defined mutation in the cystic fibrosis transmembrane regulator (CFTR) (e.g., any of the known variants of the CFTR gene, such as the delta F508 allele).

Patients will have been tested or will be tested for the CFTR gene under another protocol.

Research volunteers that are age-and race-matched as control subjects.

EXCLUSION CRITERIA:

Patients who are less than 9 years of age. Research volunteers less than 18 years of age.

Patients or research volunteers who test positive for human immunodeficiency virus (HIV) or a positive serum test for hepatitis B and/or C virus.

Patients or research volunteers who test positive for tuberculosis.

Research volunteers with pulmonary disease or infection.

Ages: 9 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with cystic fibrosis being treated with antibiotics, patients with cystic fibrosis who have not undergone antibiotic therapy, and control patients.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 1998-03-17 (Actual); Primary Completion 2006-09-07 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Serum will be analyzed for the presence of an immune response, focusing on antibodies against the virulence determinants, whilesputum will be analyzed for the immunological and genetic presence of the virulence determinants. | End of Study
  serum will be analyzed for the presence of an immune response, focusing on antibodies against the virulence determinants, whilesputum will be analyzed for the immunological and genetic presence of the virulence determinants.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Moss, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Finck-Barbancon V, Goranson J, Zhu L, Sawa T, Wiener-Kronish JP, Fleiszig SM, Wu C, Mende-Mueller L, Frank DW. ExoU expression by Pseudomonas aeruginosa correlates with acute cytotoxicity and epithelial injury. Mol Microbiol. 1997 Aug;25(3):547-57. doi: 10.1046/j.1365-2958.1997.4891851.x. PMID 9302017
- [Background] Fu H, Coburn J, Collier RJ. The eukaryotic host factor that activates exoenzyme S of Pseudomonas aeruginosa is a member of the 14-3-3 protein family. Proc Natl Acad Sci U S A. 1993 Mar 15;90(6):2320-4. doi: 10.1073/pnas.90.6.2320. PMID 8460141
- [Background] Frank DW. The exoenzyme S regulon of Pseudomonas aeruginosa. Mol Microbiol. 1997 Nov;26(4):621-9. doi: 10.1046/j.1365-2958.1997.6251991.x. PMID 9427393
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1998-H-0062.html